CLINICAL TRIAL: NCT01629134
Title: Postmarket Study of JUVÉDERM VOLBELLA™ With Lidocaine in the Lips
Status: Completed | Type: Observational
Sponsor: Allergan Medical (Industry)
Responsible Party: Sponsor
Organization: Allergan (Industry)
Other Study IDs: MAF/AGN/MED/FIL/019
Record Dates: First submitted 2012-06-25; First posted 2012-06-27 (Estimated); Results first posted 2013-05-14 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2014-10

CONDITIONS: Lip Augmentation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Volbella: Subjects treated with JUVÉDERM VOLBELLA™ according to the physician's experience and Directions for Use
  Interventions: Device: Crosslinked hyaluronic acid gel

INTERVENTIONS:
Device: Crosslinked hyaluronic acid gel — All treatments are carried out according to the physician's experience and the Directions for Use
  Other Names: JUVÉDERM VOLBELLA™

SUMMARY:
A prospective, multicenter postmarket study of the use of JUVÉDERM VOLBELLA™ with Lidocaine in the lips.

ELIGIBILITY:
Inclusion Criteria:

* Desire and willingness for correction of asymmetry or volume enhancement of his/her lips
* Females and males ≥ 18 years of age
* Have established a realistic treatment goal that the Physician agrees is achievable, i.e., have realistic expectations of aesthetic results

Exclusion Criteria:

* Not fulfilling the standard prescribing criteria for JUVÉDERM VOLBELLA™ with Lidocaine as detailed in the Directions for Use
* Have a condition or be in a situation that, in the Physician's opinion, may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers desiring lip augmentation
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2012-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Allergan Medical
Locations (1):
- Düsseldorf, North Rhine-Westphalia, Germany

REFERENCES:
- [Result] Philipp-Dormston WG, Hilton S, Nathan M. A prospective, open-label, multicenter, observational, postmarket study of the use of a 15 mg/mL hyaluronic acid dermal filler in the lips. J Cosmet Dermatol. 2014 Jun;13(2):125-34. doi: 10.1111/jocd.12085. PMID 24910276

RESULTS

PARTICIPANT FLOW:
Groups:
- Volbella: Subjects treated with JUVÉDERM VOLBELLA™ according to the physician's experience and Directions for Use
  Crosslinked hyaluronic acid gel : All treatments are carried out according to the physician's experience and the Directions for Use
Period: Overall Study
Arm/Group | Volbella
Started | 62
Completed | 62
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Volbella
Number analyzed (Participants) | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 59
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.7 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 7
Region of Enrollment [Number; unit: participants]
  Germany | 62

OUTCOME MEASURES:

1. Primary Outcome: Subject Rating of the Natural Look and Feel of the Lips
Description: Percentage of subjects rating the look and feel of their lips as being extremely natural, very natural, slightly natural, and not natural.
Time Frame: 4 weeks
Population: All subjects who met the criteria and treatment was initiated
Measure: Number; unit: Percentage of subjects
Arm/Group | Volbella
Number analyzed (Participants) | 59
Percentage of subjects
  Extremely natural | 52.5
  Very natural | 35.6
  Slightly natural | 11.9
  Not natural | 0

2. Primary Outcome: Injector Rating of the Natural Look and Feel of the Lips
Description: Percentage of injectors who rated the look and feel of subjects' lips as being extremely natural, very natural, slightly natural, and not natural.
Time Frame: 4 weeks
Population: All subjects who met the criteria and treatment was initiated
Measure: Number; unit: Percentage of subjects
Arm/Group | Volbella
Number analyzed (Participants) | 61
Percentage of subjects
  Extremely natural | 45.9
  Very natural | 54.1
  Slightly natural | 0
  Not natural | 0

3. Secondary Outcome: Bruising of the Lips
Description: Injector assessment of whether there was none, little, some, moderate, or considerable bruising in subjects' lips
Time Frame: 15 minutes after injection
Population: All subjects who met the criteria and treatment was initiated
Measure: Number; unit: Percentage of subjects
Arm/Group | Volbella
Number analyzed (Participants) | 62
Percentage of subjects
  None | 85.5
  Little | 12.9
  Some | 1.6
  Moderate | 0
  Considerable | 0

4. Secondary Outcome: Swelling of the Lips
Description: Injector assessment of whether there was none, little, some, moderate, or considerable swelling in subjects' lips
Time Frame: 15 minutes after injection
Population: All subjects who met the criteria and treatment was initiated
Measure: Number; unit: Percentage of subjects
Arm/Group | Volbella
Number analyzed (Participants) | 62
Percentage of subjects
  None | 38.7
  Little | 53.2
  Some | 8.1
  Moderate | 0
  Considerable | 0

5. Secondary Outcome: Ease of Injection
Description: Injectors rated the ease of injection on a scale ranging from 0 (Very easy) to 10 (Extremely difficult)
Time Frame: 15 minutes after injection
Population: All subjects who met the criteria and treatment was initiated
Measure: Number; unit: Percentage of subjects
Arm/Group | Volbella
Number analyzed (Participants) | 62
Percentage of subjects
  Score of 0 | 54.8
  Score of 1 | 45.2

6. Secondary Outcome: Malleability of Product
Description: Injectors rated the malleability on a scale ranging from 0 (Extremely malleable/Not hard to mold) to 10 (Not malleable/Hard to mold)
Time Frame: 15 minutes after injection
Population: All subjects who met the criteria and treatment was initiated
Measure: Number; unit: Percentage of subjects
Arm/Group | Volbella
Number analyzed (Participants) | 62
Percentage of subjects
  Score of 0 | 45.2
  Score of 1 | 54.8

7. Secondary Outcome: Need for Massage
Description: Injectors rated whether none/minimal, a little, some, or a lot of massage was required to optimize placement of VOLBELLA
Time Frame: 15 minutes after injection
Population: All subjects who met the criteria and treatment was initiated
Measure: Number; unit: Percentage of subjects
Arm/Group | Volbella
Number analyzed (Participants) | 62
Percentage of subjects
  None/minimal | 41.9
  A little | 58.1
  Some | 0
  A lot | 0

8. Secondary Outcome: Return to Social Engagement
Description: Time to return to normal daily activities
Time Frame: 4 weeks
Population: All subjects who met the criteria and treatment was initiated
Measure: Number; unit: Percentage of subjects
Arm/Group | Volbella
Number analyzed (Participants) | 61
Percentage of subjects
  < 1 Day (same day) | 62.3
  1 Day (next day) | 19.7
  2-3 Days | 9.8
  4-5 Days | 8.2
  > 6 Days | 0

9. Secondary Outcome: Comparative Rating With Previous Treatment
Description: Subject rating of lip improvement with VOLBELLA compared with previous lip enhancement treatments as significantly better, somewhat better, no difference, somewhat worse, or significantly worse
Time Frame: 15 minutes after injection
Population: All subjects who met the criteria and treatment was initiated
Measure: Number; unit: Percentage of subjects
Arm/Group | Volbella
Number analyzed (Participants) | 13
Percentage of subjects
  Significantly better | 46.2
  Somewhat better | 53.8
  No difference | 0
  Somewhat worse | 0
  Significantly worse | 0

10. Secondary Outcome: Rating of Injection Discomfort
Description: The level of discomfort during treatment on a scale of 0 (no discomfort) to 10 (extreme discomfort).
Time Frame: 15 minutes after injection
Population: All subjects who met the criteria and treatment was initiated
Measure: Mean (Standard Deviation); unit: scale score
Arm/Group | Volbella
Number analyzed (Participants) | 58
scale score | 1.3 (1.5)

ADVERSE EVENTS:
Arm/Group | Volbella
Serious Adverse Events (participants affected / at risk) | 0/62
Other Adverse Events (participants affected / at risk) | 0/62

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No